CLINICAL TRIAL: NCT01858662
Title: Randomised Phase 2 Study Comparing Pathological Responses Observed on Colorectal Cancer Metastases Resected After Preoperative Treatment Combining Cetuximab With FOLFOX or FOLFIRI in RAS and B-RAF WT Tumors
Brief Title: Study Comparing Pathological Responses Observed on Colorectal Cancer Metastases Resected After Preoperative Treatment Combining Cetuximab With FOLFOX or FOLFIRI in RAS and B-RAF WT Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to poor recrutment
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Grand Hôpital de Charleroi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CET-ONCO2012; 2012-005249-19 (EudraCT Number)
Record Dates: First submitted 2013-05-07; First posted 2013-05-21 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic colorectal cancer; Liver; cetuximab; Pathological response
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Leucovorin; Oxaliplatin; Irinotecan; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oxaliplatin +leucovorin L+5FU+ cetuximab (Active Comparator): oxaliplatin +leucovorinL+5-Fluorouracile +cetuximab+'Metastases Resection ( multiple steep surgery possible)
  Interventions: Procedure: Metastases Resection ( multiple steep surgery possible); Drug: 5-Fluorouracile; Drug: leucovorin L; Drug: Oxaliplatin; Drug: Cetuximab
- Irinotecan+ + leucovorinL +5-Fluorouracil +cetuximab (Active Comparator): Irinotecan+ + leucovorinL +5-Fluorouracile + cetuximab +'Metastases Resection ( multiple steep surgery possible)
  Interventions: Procedure: Metastases Resection ( multiple steep surgery possible); Drug: 5-Fluorouracile; Drug: leucovorin L; Drug: Irinotecan; Drug: Cetuximab

INTERVENTIONS:
Procedure: Metastases Resection ( multiple steep surgery possible) — Metastases resection will be process by surgery, after a randomized chemotherapy (FOLFOX or FOLFIRI) + Target therapy (Cetuximab). The surgery will allow to compare the pathological response on the resected metastases by the chemotherapy + target therapy type.
Drug: 5-Fluorouracile — 5-FU bolus 400 mg/m2, IV bolus every 2 weeks 5-FU continuous infusion 2400 mg/m2, 46-hour cont. IV infusion every 2 weeks
  Other Names: 5FU
Drug: leucovorin L — Leucovorin L (levoleucovorin) 200 mg/m2 (or folinic acid 400 mg/m²) in 250 ml glucose 5%, 2-hour IV infusion
  Other Names: elvorine; isovorin
Drug: Oxaliplatin — Oxaliplatin 85 mg/m² in 150 ml NaCl 0.9%, 2-hour IV infusion every 2 weeks
  Other Names: Eloxatin
  Arms: oxaliplatin +leucovorin L+5FU+ cetuximab
Drug: Irinotecan — Irinotecan 180 mg/m² in 150 ml NaCl 0.9%, 1.30-hour IV infusion every 2 weeks
  Other Names: Campto; Irinosin
  Arms: Irinotecan+ + leucovorinL +5-Fluorouracil +cetuximab
Drug: Cetuximab — Cetuximab 400 mg/m² in 100 ml NaCl 0.9% 2-hour IV infusion for 1rst cycle and after the 1rst cycle 250 mg/m² in 100 ml NaCl 0.9% 1-hour IV infusion
  Other Names: erbitux

SUMMARY:
To analyze the pathological tumor response on resected colorectal cancer metastases after preoperative treatment with cetuximab combined with FOLFOX or FOLFIRI regimen in a prospective cohort (RAS and B-RAF WT tumors) and to correlate this response with patient's outcome.

DETAILED DESCRIPTION:
This is a phase II , openlabel, randomized study in patients with confirmed diagnosis of potentially or borderline resectable metastatic colorectal adenocarcinoma (RAS and B-RAF WT tumors ), who have not received prior chemotherapy for their metastatic disease.

The study is designed to compare pathological responses observed after pre-operative chemotherapy cetuximab with FOLFOX or FOLFIRI.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male patients with at least 18 years at the time the informed consent is signed
2. ECOG performance status 0 or 1
3. Histological or cytological confirmed diagnostic of adenocarcinoma of the colon or rectum, with or without primary tumour in situ. Wild-type RAS and B-RAF tumor status.
4. Patients with potentially resectable metastatic disease at diagnosis and for whom a chemotherapy first in a curative intent is recommended . Resectability could be planed in one or multiple stage if indicated. As commonly admitted, resectability means the surgical clearance (+/- radiofrequency ablation) of all detectable (liver) lesions with tumor-free margins and compatible with an adequate hepatic reserve. Practically, bilateral tumor location, number and location of lesions, and inadequate hepatic reserve remain the main decisional factors.
5. Partial and minor resection of metastatic disease is allowed within 3 months before inclusion if patient has never received chemotherapy for mCRC.
6. Extra hepatic metastatic location is limited to 1 site.
7. Patients may have received adjuvant chemotherapy or (neo-) adjuvant chemo-radiotherapy to the pelvis, provided the last dose of chemotherapy was administered at least 6 months prior to inclusion (12 months for oxaliplatin). Previous radiotherapy to the pelvis is not an exclusion criterion.
8. Adequate haematological, renal and hepatic function as follows:

   Haematological:

   haemoglobin >9g/dl Neutrophils > 1.5 x 109/L Platelets > 100 x 109/L

   Renal:

   Creatinine< 1.5 x ULN (Upper Limit of Normal)

   Hepatic:

   Bilirubin < or equal 1.5 X ULN AST (Aspartate Aminotransferase),and ALT (Alanine Aminotransferase)< or equal 5 x ULN, Phos Alc< or equal 5 x ULN
9. Female patients must either be postmenopausal, sterile (surgically or radiation- or chemically-induced), or if sexually active using an acceptable method of contraception.
10. Male patients must be surgically sterile or if sexually active and having a pre-menopausal partner must be using an acceptable method of contraception.
11. Life expectancy of at least 3 months without any active treatment.

Exclusion Criteria:

* 1.Definitively non resectable mCRC at diagnosis
* 2.Prior chemotherapy or systemic therapy for mCRC. Adjuvant chemotherapy for colorectal cancer is not an exclusion criterion provided that it was completed more than 6 months prior to inclusion. Oxaliplatin-based chemotherapy must be completed more than 1 year prior to inclusion.
* 3.Prior utilization of cetuximab, panitumumab (or other anti-EGFR (epidermal growth factor receptor)therapy).
* 4.Previous radiotherapy delivered to the upper abdomen.
* 5 Non mesurable disease( RECIST 1.1 criteria)
* 6.Evidence of ascites, cirrhosis, portal hypertension, main portal venous tumour involvement or thrombosis as determined by clinical or radiologic assessment.
* 7.Prior major liver resection: remnant liver < 50% of the initial liver volume.
* 8.Non-malignant disease that would render the patient unsuitable for treatment according to this protocol.
* 9.Concurrent central nervous systems metastases
* 10.Peripheric neuropathy ≥ grade 2.
* 11.Interstitial lung disease
* 12.Pregnant or breast feeding.
* 13.The patient has previous or concomitant malignancies, except: Invasive malignancies in remission for more than 5 years and non melanoma skin cancer or carcinoma in situ of the cervix.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Major Pathological Response Rate | Average 3 months (after resection of metastases)
  Major pathological response rate (MPRR) is defined as the proportion of patients presenting a major pathological response. Pathologic response will be evaluated according the Rubbia-Brandt Tumor Regression Grade classification .For patients with multiple colorectal metastases the global pathological response will be categorized based on the mean TRG of all metastases.: a major response is defined as a mean TRG < 3, a partial response is defined for patient presenting a mean TRG ≥3 and <4, and a no response for patient with a mean TRG ≥4.

SECONDARY OUTCOMES:
progression free survival | at 6 months and at 12 months after randomization
  -Progression Free Survival (PFS) is defined as the time from randomization to the time of first event (relapse of the original mCRC, development of a new colorectal cancer or death due to any cause). Patients without any such event at the time of data analysis will be censored at the last date they were known to be event-free. PFS analysis will be based on tumour assessments and survival follow-up assessments.
Overall survival | At the end of the study
  The overall survival will be analyzed at the end of study (3 year of recruitment and one year of follow-up).
Clinical response rate | at time of surgery -
  Clinical response rate at time of surgery: Clinical tumour response will be measured according to the RECIST 1.1 criteria
Metabolic response rate | At time of surgery - average 3 months
  Metabolic response rate at time of surgery (in selected centres only, optional): Metabolic tumour response will be measured according to the EORTC criteria . PET-Scan evaluation remains optional to selected centres only.
post operative complications | one month after surgery
  . Severe pre- or postoperative complications within 30 days of surgery:
  * surgery-associated bleeding requiring replacement with > 4 units of erythrocyte concentrates,
  * wound infection,
  * intra-abdominal infection,
  * severe sepsis (American College of Chest physicians/Society of Critical Care Medicine, 1992),
  * impaired wound healing,
  * subphrenic or perihepatic abscess requiring drainage during hospital stay or within 30 days after the operation,
  * re-laparotomy connected with the resection,
  * a biliary fistula for more than 10 days with a discharge of > 100 mL/day,
  * transient liver failure (bilirubin > 10 mg/dL lasting > 3 days),
  * renal failure requiring dialysis,
  * respiratory failure with renewed necessary mechanical ventilation, venous thromboembolism,
  * cardiac failure,
  * death of the patient as a result of the operation.
Curative resection rate | At time of surgery
  Curative resection rate (R0 resection) is defined by the surgical clearance (+/- radiofrequency ablation) of all detectable hepatic lesions with tumor-free margins at histo-pathological evaluation.
Chemotherapy-associated hepatotoxicity: | at time of surgery
  Systemic neo-adjuvant chemotherapy in mCRC frequently causes morphological lesions involving hepatic microvasculature . Sinusoidal obstruction, complicated by perisinusoidal fibrosis and veno-occlusive lesion of the non tumoral liver, should be included in the list of the adverse side-effects of colorectal systemic chemotherapy, in particular related to the use of oxaliplatin.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Van den Eynde, MD, Principal Investigator — Cliniques universitaires Saint-Luc - UCL; Javier Carrasco, MD PhD, Principal Investigator — Grand Hôpital de Charleroi
Locations (7):
- Belgium (7):
  - Cliniques universitaires Saint-Luc - UCL, Brussels, Brussels Capital
  - Grand Hôpital de Charleroi, Charleroi, Hainaut
  - clinique Saint Luc, Bouge
  - Centre Hospitalier Jolimont Lobbes, La Louvière
  - CHU liège (Sart Timan), Liège
  - Clinique Saint Pierre Ottignies, Ottignies
  - CHU-UCL Dinant-Godinne, Yvoir

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Thun MJ. Cancer statistics, 2009. CA Cancer J Clin. 2009 Jul-Aug;59(4):225-49. doi: 10.3322/caac.20006. Epub 2009 May 27. PMID 19474385
- [Background] Jamison RL, Donohue JH, Nagorney DM, Rosen CB, Harmsen WS, Ilstrup DM. Hepatic resection for metastatic colorectal cancer results in cure for some patients. Arch Surg. 1997 May;132(5):505-10; discussion 511. doi: 10.1001/archsurg.1997.01430290051008. PMID 9161393
- [Background] Nordlinger B, Guiguet M, Vaillant JC, Balladur P, Boudjema K, Bachellier P, Jaeck D. Surgical resection of colorectal carcinoma metastases to the liver. A prognostic scoring system to improve case selection, based on 1568 patients. Association Francaise de Chirurgie. Cancer. 1996 Apr 1;77(7):1254-62. PMID 8608500
- [Background] Rees M, Tekkis PP, Welsh FK, O'Rourke T, John TG. Evaluation of long-term survival after hepatic resection for metastatic colorectal cancer: a multifactorial model of 929 patients. Ann Surg. 2008 Jan;247(1):125-35. doi: 10.1097/SLA.0b013e31815aa2c2. PMID 18156932
- [Background] Nordlinger B, Sorbye H, Glimelius B, Poston GJ, Schlag PM, Rougier P, Bechstein WO, Primrose JN, Walpole ET, Finch-Jones M, Jaeck D, Mirza D, Parks RW, Collette L, Praet M, Bethe U, Van Cutsem E, Scheithauer W, Gruenberger T; EORTC Gastro-Intestinal Tract Cancer Group; Cancer Research UK; Arbeitsgruppe Lebermetastasen und-tumoren in der Chirurgischen Arbeitsgemeinschaft Onkologie (ALM-CAO); Australasian Gastro-Intestinal Trials Group (AGITG); Federation Francophone de Cancerologie Digestive (FFCD). Perioperative chemotherapy with FOLFOX4 and surgery versus surgery alone for resectable liver metastases from colorectal cancer (EORTC Intergroup trial 40983): a randomised controlled trial. Lancet. 2008 Mar 22;371(9617):1007-16. doi: 10.1016/S0140-6736(08)60455-9. PMID 18358928
- [Background] Hurwitz H, Fehrenbacher L, Novotny W, Cartwright T, Hainsworth J, Heim W, Berlin J, Baron A, Griffing S, Holmgren E, Ferrara N, Fyfe G, Rogers B, Ross R, Kabbinavar F. Bevacizumab plus irinotecan, fluorouracil, and leucovorin for metastatic colorectal cancer. N Engl J Med. 2004 Jun 3;350(23):2335-42. doi: 10.1056/NEJMoa032691. PMID 15175435
- [Background] Saltz LB, Clarke S, Diaz-Rubio E, Scheithauer W, Figer A, Wong R, Koski S, Lichinitser M, Yang TS, Rivera F, Couture F, Sirzen F, Cassidy J. Bevacizumab in combination with oxaliplatin-based chemotherapy as first-line therapy in metastatic colorectal cancer: a randomized phase III study. J Clin Oncol. 2008 Apr 20;26(12):2013-9. doi: 10.1200/JCO.2007.14.9930. PMID 18421054
- [Background] Van Cutsem E, Kohne CH, Lang I, Folprecht G, Nowacki MP, Cascinu S, Shchepotin I, Maurel J, Cunningham D, Tejpar S, Schlichting M, Zubel A, Celik I, Rougier P, Ciardiello F. Cetuximab plus irinotecan, fluorouracil, and leucovorin as first-line treatment for metastatic colorectal cancer: updated analysis of overall survival according to tumor KRAS and BRAF mutation status. J Clin Oncol. 2011 May 20;29(15):2011-9. doi: 10.1200/JCO.2010.33.5091. Epub 2011 Apr 18. PMID 21502544
- [Background] Bokemeyer C, Van Cutsem E, Rougier P, Ciardiello F, Heeger S, Schlichting M, Celik I, Kohne CH. Addition of cetuximab to chemotherapy as first-line treatment for KRAS wild-type metastatic colorectal cancer: pooled analysis of the CRYSTAL and OPUS randomised clinical trials. Eur J Cancer. 2012 Jul;48(10):1466-75. doi: 10.1016/j.ejca.2012.02.057. Epub 2012 Mar 23. PMID 22446022
- [Background] Douillard JY, Siena S, Cassidy J, Tabernero J, Burkes R, Barugel M, Humblet Y, Bodoky G, Cunningham D, Jassem J, Rivera F, Kocakova I, Ruff P, Blasinska-Morawiec M, Smakal M, Canon JL, Rother M, Oliner KS, Wolf M, Gansert J. Randomized, phase III trial of panitumumab with infusional fluorouracil, leucovorin, and oxaliplatin (FOLFOX4) versus FOLFOX4 alone as first-line treatment in patients with previously untreated metastatic colorectal cancer: the PRIME study. J Clin Oncol. 2010 Nov 1;28(31):4697-705. doi: 10.1200/JCO.2009.27.4860. Epub 2010 Oct 4. PMID 20921465
- [Background] Khatri VP, Chee KG, Petrelli NJ. Modern multimodality approach to hepatic colorectal metastases: solutions and controversies. Surg Oncol. 2007 Jul;16(1):71-83. doi: 10.1016/j.suronc.2007.05.001. Epub 2007 May 29. PMID 17532622
- [Background] de Gramont A, Tournigand C, Andre T, Larsen AK, Louvet C. Adjuvant therapy for stage II and III colorectal cancer. Semin Oncol. 2007 Apr;34(2 Suppl 1):S37-40. doi: 10.1053/j.seminoncol.2007.01.004. PMID 17449351
- [Background] Andre T, Boni C, Mounedji-Boudiaf L, Navarro M, Tabernero J, Hickish T, Topham C, Zaninelli M, Clingan P, Bridgewater J, Tabah-Fisch I, de Gramont A; Multicenter International Study of Oxaliplatin/5-Fluorouracil/Leucovorin in the Adjuvant Treatment of Colon Cancer (MOSAIC) Investigators. Oxaliplatin, fluorouracil, and leucovorin as adjuvant treatment for colon cancer. N Engl J Med. 2004 Jun 3;350(23):2343-51. doi: 10.1056/NEJMoa032709. PMID 15175436
- [Background] Gruenberger B, Tamandl D, Schueller J, Scheithauer W, Zielinski C, Herbst F, Gruenberger T. Bevacizumab, capecitabine, and oxaliplatin as neoadjuvant therapy for patients with potentially curable metastatic colorectal cancer. J Clin Oncol. 2008 Apr 10;26(11):1830-5. doi: 10.1200/JCO.2007.13.7679. PMID 18398148
- [Background] Klinger M, Tamandl D, Eipeldauer S, Hacker S, Herberger B, Kaczirek K, Dorfmeister M, Gruenberger B, Gruenberger T. Bevacizumab improves pathological response of colorectal cancer liver metastases treated with XELOX/FOLFOX. Ann Surg Oncol. 2010 Aug;17(8):2059-65. doi: 10.1245/s10434-010-0972-9. Epub 2010 Feb 23. PMID 20177795
- [Background] Folprecht G, Gruenberger T, Bechstein WO, Raab HR, Lordick F, Hartmann JT, Lang H, Frilling A, Stoehlmacher J, Weitz J, Konopke R, Stroszczynski C, Liersch T, Ockert D, Herrmann T, Goekkurt E, Parisi F, Kohne CH. Tumour response and secondary resectability of colorectal liver metastases following neoadjuvant chemotherapy with cetuximab: the CELIM randomised phase 2 trial. Lancet Oncol. 2010 Jan;11(1):38-47. doi: 10.1016/S1470-2045(09)70330-4. Epub 2009 Nov 26. PMID 19942479
- [Background] Maughan TS, Adams RA, Smith CG, Meade AM, Seymour MT, Wilson RH, Idziaszczyk S, Harris R, Fisher D, Kenny SL, Kay E, Mitchell JK, Madi A, Jasani B, James MD, Bridgewater J, Kennedy MJ, Claes B, Lambrechts D, Kaplan R, Cheadle JP; MRC COIN Trial Investigators. Addition of cetuximab to oxaliplatin-based first-line combination chemotherapy for treatment of advanced colorectal cancer: results of the randomised phase 3 MRC COIN trial. Lancet. 2011 Jun 18;377(9783):2103-14. doi: 10.1016/S0140-6736(11)60613-2. Epub 2011 Jun 5. PMID 21641636
- [Background] Tveit KM, Guren T, Glimelius B, Pfeiffer P, Sorbye H, Pyrhonen S, Sigurdsson F, Kure E, Ikdahl T, Skovlund E, Fokstuen T, Hansen F, Hofsli E, Birkemeyer E, Johnsson A, Starkhammar H, Yilmaz MK, Keldsen N, Erdal AB, Dajani O, Dahl O, Christoffersen T. Phase III trial of cetuximab with continuous or intermittent fluorouracil, leucovorin, and oxaliplatin (Nordic FLOX) versus FLOX alone in first-line treatment of metastatic colorectal cancer: the NORDIC-VII study. J Clin Oncol. 2012 May 20;30(15):1755-62. doi: 10.1200/JCO.2011.38.0915. Epub 2012 Apr 2. PMID 22473155
- [Background] Gralow JR, Burstein HJ, Wood W, Hortobagyi GN, Gianni L, von Minckwitz G, Buzdar AU, Smith IE, Symmans WF, Singh B, Winer EP. Preoperative therapy in invasive breast cancer: pathologic assessment and systemic therapy issues in operable disease. J Clin Oncol. 2008 Feb 10;26(5):814-9. doi: 10.1200/JCO.2007.15.3510. PMID 18258991
- [Background] Mandard AM, Dalibard F, Mandard JC, Marnay J, Henry-Amar M, Petiot JF, Roussel A, Jacob JH, Segol P, Samama G, et al. Pathologic assessment of tumor regression after preoperative chemoradiotherapy of esophageal carcinoma. Clinicopathologic correlations. Cancer. 1994 Jun 1;73(11):2680-6. doi: 10.1002/1097-0142(19940601)73:113.0.co;2-c. PMID 8194005
- [Background] Swisher SG, Hofstetter W, Wu TT, Correa AM, Ajani JA, Komaki RR, Chirieac L, Hunt KK, Liao Z, Phan A, Rice DC, Vaporciyan AA, Walsh GL, Roth JA. Proposed revision of the esophageal cancer staging system to accommodate pathologic response (pP) following preoperative chemoradiation (CRT). Ann Surg. 2005 May;241(5):810-7; discussion 817-20. doi: 10.1097/01.sla.0000161983.82345.85. PMID 15849517
- [Background] Ajani JA, Mansfield PF, Crane CH, Wu TT, Lunagomez S, Lynch PM, Janjan N, Feig B, Faust J, Yao JC, Nivers R, Morris J, Pisters PW. Paclitaxel-based chemoradiotherapy in localized gastric carcinoma: degree of pathologic response and not clinical parameters dictated patient outcome. J Clin Oncol. 2005 Feb 20;23(6):1237-44. doi: 10.1200/JCO.2005.01.305. PMID 15718321
- [Background] Rodel C, Martus P, Papadoupolos T, Fuzesi L, Klimpfinger M, Fietkau R, Liersch T, Hohenberger W, Raab R, Sauer R, Wittekind C. Prognostic significance of tumor regression after preoperative chemoradiotherapy for rectal cancer. J Clin Oncol. 2005 Dec 1;23(34):8688-96. doi: 10.1200/JCO.2005.02.1329. Epub 2005 Oct 24. PMID 16246976
- [Background] Bouzourene H, Bosman FT, Seelentag W, Matter M, Coucke P. Importance of tumor regression assessment in predicting the outcome in patients with locally advanced rectal carcinoma who are treated with preoperative radiotherapy. Cancer. 2002 Feb 15;94(4):1121-30. PMID 11920483
- [Background] Rubbia-Brandt L, Giostra E, Brezault C, Roth AD, Andres A, Audard V, Sartoretti P, Dousset B, Majno PE, Soubrane O, Chaussade S, Mentha G, Terris B. Importance of histological tumor response assessment in predicting the outcome in patients with colorectal liver metastases treated with neo-adjuvant chemotherapy followed by liver surgery. Ann Oncol. 2007 Feb;18(2):299-304. doi: 10.1093/annonc/mdl386. Epub 2006 Oct 23. PMID 17060484
- [Background] Ribero D, Wang H, Donadon M, Zorzi D, Thomas MB, Eng C, Chang DZ, Curley SA, Abdalla EK, Ellis LM, Vauthey JN. Bevacizumab improves pathologic response and protects against hepatic injury in patients treated with oxaliplatin-based chemotherapy for colorectal liver metastases. Cancer. 2007 Dec 15;110(12):2761-7. doi: 10.1002/cncr.23099. PMID 17960603
- [Background] Blazer DG 3rd, Kishi Y, Maru DM, Kopetz S, Chun YS, Overman MJ, Fogelman D, Eng C, Chang DZ, Wang H, Zorzi D, Ribero D, Ellis LM, Glover KY, Wolff RA, Curley SA, Abdalla EK, Vauthey JN. Pathologic response to preoperative chemotherapy: a new outcome end point after resection of hepatic colorectal metastases. J Clin Oncol. 2008 Nov 20;26(33):5344-51. doi: 10.1200/JCO.2008.17.5299. Epub 2008 Oct 20. PMID 18936472
- [Background] Maru DM, Kopetz S, Boonsirikamchai P, Agarwal A, Chun YS, Wang H, Abdalla EK, Kaur H, Charnsangavej C, Vauthey JN, Loyer EM. Tumor thickness at the tumor-normal interface: a novel pathologic indicator of chemotherapy response in hepatic colorectal metastases. Am J Surg Pathol. 2010 Sep;34(9):1287-94. doi: 10.1097/PAS.0b013e3181eb2f7b. PMID 20697255
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Young H, Baum R, Cremerius U, Herholz K, Hoekstra O, Lammertsma AA, Pruim J, Price P. Measurement of clinical and subclinical tumour response using [18F]-fluorodeoxyglucose and positron emission tomography: review and 1999 EORTC recommendations. European Organization for Research and Treatment of Cancer (EORTC) PET Study Group. Eur J Cancer. 1999 Dec;35(13):1773-82. doi: 10.1016/s0959-8049(99)00229-4. PMID 10673991
- [Background] Rubbia-Brandt L, Audard V, Sartoretti P, Roth AD, Brezault C, Le Charpentier M, Dousset B, Morel P, Soubrane O, Chaussade S, Mentha G, Terris B. Severe hepatic sinusoidal obstruction associated with oxaliplatin-based chemotherapy in patients with metastatic colorectal cancer. Ann Oncol. 2004 Mar;15(3):460-6. doi: 10.1093/annonc/mdh095. PMID 14998849
- [Background] Galon J, Costes A, Sanchez-Cabo F, Kirilovsky A, Mlecnik B, Lagorce-Pages C, Tosolini M, Camus M, Berger A, Wind P, Zinzindohoue F, Bruneval P, Cugnenc PH, Trajanoski Z, Fridman WH, Pages F. Type, density, and location of immune cells within human colorectal tumors predict clinical outcome. Science. 2006 Sep 29;313(5795):1960-4. doi: 10.1126/science.1129139. PMID 17008531
- [Background] Galon J, Fridman WH, Pages F. The adaptive immunologic microenvironment in colorectal cancer: a novel perspective. Cancer Res. 2007 Mar 1;67(5):1883-6. doi: 10.1158/0008-5472.CAN-06-4806. PMID 17332313
- [Background] Mlecnik B, Tosolini M, Kirilovsky A, Berger A, Bindea G, Meatchi T, Bruneval P, Trajanoski Z, Fridman WH, Pages F, Galon J. Histopathologic-based prognostic factors of colorectal cancers are associated with the state of the local immune reaction. J Clin Oncol. 2011 Feb 20;29(6):610-8. doi: 10.1200/JCO.2010.30.5425. Epub 2011 Jan 18. PMID 21245428
- [Background] Pages F, Berger A, Camus M, Sanchez-Cabo F, Costes A, Molidor R, Mlecnik B, Kirilovsky A, Nilsson M, Damotte D, Meatchi T, Bruneval P, Cugnenc PH, Trajanoski Z, Fridman WH, Galon J. Effector memory T cells, early metastasis, and survival in colorectal cancer. N Engl J Med. 2005 Dec 22;353(25):2654-66. doi: 10.1056/NEJMoa051424. PMID 16371631
- [Background] Pages F, Kirilovsky A, Mlecnik B, Asslaber M, Tosolini M, Bindea G, Lagorce C, Wind P, Marliot F, Bruneval P, Zatloukal K, Trajanoski Z, Berger A, Fridman WH, Galon J. In situ cytotoxic and memory T cells predict outcome in patients with early-stage colorectal cancer. J Clin Oncol. 2009 Dec 10;27(35):5944-51. doi: 10.1200/JCO.2008.19.6147. Epub 2009 Oct 26. PMID 19858404
- [Background] Butterfield LH, Disis ML, Fox BA, Lee PP, Khleif SN, Thurin M, Trinchieri G, Wang E, Wigginton J, Chaussabel D, Coukos G, Dhodapkar M, Hakansson L, Janetzki S, Kleen TO, Kirkwood JM, Maccalli C, Maecker H, Maio M, Malyguine A, Masucci G, Palucka AK, Potter DM, Ribas A, Rivoltini L, Schendel D, Seliger B, Selvan S, Slingluff CL Jr, Stroncek DF, Streicher H, Wu X, Zeskind B, Zhao Y, Zocca MB, Zwierzina H, Marincola FM. A systematic approach to biomarker discovery; preamble to "the iSBTc-FDA taskforce on immunotherapy biomarkers". J Transl Med. 2008 Dec 23;6:81. doi: 10.1186/1479-5876-6-81. PMID 19105846
- [Background] Butterfield LH, Palucka AK, Britten CM, Dhodapkar MV, Hakansson L, Janetzki S, Kawakami Y, Kleen TO, Lee PP, Maccalli C, Maecker HT, Maino VC, Maio M, Malyguine A, Masucci G, Pawelec G, Potter DM, Rivoltini L, Salazar LG, Schendel DJ, Slingluff CL Jr, Song W, Stroncek DF, Tahara H, Thurin M, Trinchieri G, van Der Burg SH, Whiteside TL, Wigginton JM, Marincola F, Khleif S, Fox BA, Disis ML. Recommendations from the iSBTc-SITC/FDA/NCI Workshop on Immunotherapy Biomarkers. Clin Cancer Res. 2011 May 15;17(10):3064-76. doi: 10.1158/1078-0432.CCR-10-2234. Epub 2011 May 10. PMID 21558394
- [Background] Tahara H, Sato M, Thurin M, Wang E, Butterfield LH, Disis ML, Fox BA, Lee PP, Khleif SN, Wigginton JM, Ambs S, Akutsu Y, Chaussabel D, Doki Y, Eremin O, Fridman WH, Hirohashi Y, Imai K, Jacobson J, Jinushi M, Kanamoto A, Kashani-Sabet M, Kato K, Kawakami Y, Kirkwood JM, Kleen TO, Lehmann PV, Liotta L, Lotze MT, Maio M, Malyguine A, Masucci G, Matsubara H, Mayrand-Chung S, Nakamura K, Nishikawa H, Palucka AK, Petricoin EF, Pos Z, Ribas A, Rivoltini L, Sato N, Shiku H, Slingluff CL, Streicher H, Stroncek DF, Takeuchi H, Toyota M, Wada H, Wu X, Wulfkuhle J, Yaguchi T, Zeskind B, Zhao Y, Zocca MB, Marincola FM. Emerging concepts in biomarker discovery; the US-Japan Workshop on Immunological Molecular Markers in Oncology. J Transl Med. 2009 Jun 17;7:45. doi: 10.1186/1479-5876-7-45. PMID 19534815
- [Background] Bindea G, Mlecnik B, Fridman WH, Pages F, Galon J. Natural immunity to cancer in humans. Curr Opin Immunol. 2010 Apr;22(2):215-22. doi: 10.1016/j.coi.2010.02.006. Epub 2010 Mar 6. PMID 20207124
- [Background] Pages F, Galon J, Dieu-Nosjean MC, Tartour E, Sautes-Fridman C, Fridman WH. Immune infiltration in human tumors: a prognostic factor that should not be ignored. Oncogene. 2010 Feb 25;29(8):1093-102. doi: 10.1038/onc.2009.416. Epub 2009 Nov 30. PMID 19946335
- [Background] Broussard EK, Disis ML. TNM staging in colorectal cancer: T is for T cell and M is for memory. J Clin Oncol. 2011 Feb 20;29(6):601-3. doi: 10.1200/JCO.2010.32.9078. Epub 2011 Jan 18. No abstract available. PMID 21245434
- [Background] Halama N, Michel S, Kloor M, Zoernig I, Benner A, Spille A, Pommerencke T, von Knebel DM, Folprecht G, Luber B, Feyen N, Martens UM, Beckhove P, Gnjatic S, Schirmacher P, Herpel E, Weitz J, Grabe N, Jaeger D. Localization and density of immune cells in the invasive margin of human colorectal cancer liver metastases are prognostic for response to chemotherapy. Cancer Res. 2011 Sep 1;71(17):5670-7. doi: 10.1158/0008-5472.CAN-11-0268. Epub 2011 Aug 16. PMID 21846824
- [Background] Camus M, Tosolini M, Mlecnik B, Pages F, Kirilovsky A, Berger A, Costes A, Bindea G, Charoentong P, Bruneval P, Trajanoski Z, Fridman WH, Galon J. Coordination of intratumoral immune reaction and human colorectal cancer recurrence. Cancer Res. 2009 Mar 15;69(6):2685-93. doi: 10.1158/0008-5472.CAN-08-2654. Epub 2009 Mar 3. PMID 19258510
- [Background] Tesniere A, Apetoh L, Ghiringhelli F, Joza N, Panaretakis T, Kepp O, Schlemmer F, Zitvogel L, Kroemer G. Immunogenic cancer cell death: a key-lock paradigm. Curr Opin Immunol. 2008 Oct;20(5):504-11. doi: 10.1016/j.coi.2008.05.007. Epub 2008 Jun 23. PMID 18573340
- [Background] Ghiringhelli F, Menard C, Puig PE, Ladoire S, Roux S, Martin F, Solary E, Le Cesne A, Zitvogel L, Chauffert B. Metronomic cyclophosphamide regimen selectively depletes CD4+CD25+ regulatory T cells and restores T and NK effector functions in end stage cancer patients. Cancer Immunol Immunother. 2007 May;56(5):641-8. doi: 10.1007/s00262-006-0225-8. Epub 2006 Sep 8. PMID 16960692
- [Background] Machiels JP, Reilly RT, Emens LA, Ercolini AM, Lei RY, Weintraub D, Okoye FI, Jaffee EM. Cyclophosphamide, doxorubicin, and paclitaxel enhance the antitumor immune response of granulocyte/macrophage-colony stimulating factor-secreting whole-cell vaccines in HER-2/neu tolerized mice. Cancer Res. 2001 May 1;61(9):3689-97. PMID 11325840
- [Background] Mlecnik B, Tosolini M, Charoentong P, Kirilovsky A, Bindea G, Berger A, Camus M, Gillard M, Bruneval P, Fridman WH, Pages F, Trajanoski Z, Galon J. Biomolecular network reconstruction identifies T-cell homing factors associated with survival in colorectal cancer. Gastroenterology. 2010 Apr;138(4):1429-40. doi: 10.1053/j.gastro.2009.10.057. Epub 2009 Nov 10. PMID 19909745
- [Background] Branford S. Chronic myeloid leukemia: molecular monitoring in clinical practice. Hematology Am Soc Hematol Educ Program. 2007:376-83. doi: 10.1182/asheducation-2007.1.376. PMID 18024654
- [Background] Campbell PJ, Stephens PJ, Pleasance ED, O'Meara S, Li H, Santarius T, Stebbings LA, Leroy C, Edkins S, Hardy C, Teague JW, Menzies A, Goodhead I, Turner DJ, Clee CM, Quail MA, Cox A, Brown C, Durbin R, Hurles ME, Edwards PA, Bignell GR, Stratton MR, Futreal PA. Identification of somatically acquired rearrangements in cancer using genome-wide massively parallel paired-end sequencing. Nat Genet. 2008 Jun;40(6):722-9. doi: 10.1038/ng.128. Epub 2008 Apr 27. PMID 18438408
- [Background] Diehl F, Schmidt K, Choti MA, Romans K, Goodman S, Li M, Thornton K, Agrawal N, Sokoll L, Szabo SA, Kinzler KW, Vogelstein B, Diaz LA Jr. Circulating mutant DNA to assess tumor dynamics. Nat Med. 2008 Sep;14(9):985-90. doi: 10.1038/nm.1789. Epub 2007 Jul 31. PMID 18670422
- [Background] Yung TK, Chan KC, Mok TS, Tong J, To KF, Lo YM. Single-molecule detection of epidermal growth factor receptor mutations in plasma by microfluidics digital PCR in non-small cell lung cancer patients. Clin Cancer Res. 2009 Mar 15;15(6):2076-84. doi: 10.1158/1078-0432.CCR-08-2622. Epub 2009 Mar 10. PMID 19276259
- [Background] Leary RJ, Kinde I, Diehl F, Schmidt K, Clouser C, Duncan C, Antipova A, Lee C, McKernan K, De La Vega FM, Kinzler KW, Vogelstein B, Diaz LA Jr, Velculescu VE. Development of personalized tumor biomarkers using massively parallel sequencing. Sci Transl Med. 2010 Feb 24;2(20):20ra14. doi: 10.1126/scitranslmed.3000702. PMID 20371490
- [Background] McBride DJ, Orpana AK, Sotiriou C, Joensuu H, Stephens PJ, Mudie LJ, Hamalainen E, Stebbings LA, Andersson LC, Flanagan AM, Durbecq V, Ignatiadis M, Kallioniemi O, Heckman CA, Alitalo K, Edgren H, Futreal PA, Stratton MR, Campbell PJ. Use of cancer-specific genomic rearrangements to quantify disease burden in plasma from patients with solid tumors. Genes Chromosomes Cancer. 2010 Nov;49(11):1062-9. doi: 10.1002/gcc.20815. PMID 20725990